CLINICAL TRIAL: NCT05099965
Title: Phase II, Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of a Modified Vaccinia Ankara (MVA)-Based Anti-Cytomegalovirus (CMV) Vaccine (Triplex®), in Adults With Both Human Immunodeficiency Virus (HIV)-1 and CMV Who Are on Potent Combination ART With Conserved Immune Function
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a Modified Vaccinia Ankara (MVA)-Based Anti-Cytomegalovirus (CMV) Vaccine (Triplex®)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5355
Record Dates: First submitted 2021-09-01; First posted 2021-10-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Cytomegalovirus Infections; HIV Infections; Vaccine
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaccine Group (Active Comparator): 60 participants will receive CMV-MVA Triplex® containing 5 x 108 plaque-forming unit (pfu) ±0.5 x 108 pfu of MVA Vaccine Encoding CMV Antigens by intramuscular (IM) deltoid injections.
  Interventions: Biological: CMV-MVA Triplex
- Placebo Group (Placebo Comparator): 30 participants will receive a volume of placebo (7.5% Lactose in phosphate-buffered saline [PBS]) that matches the volume of the active vaccine injection by IM deltoid injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CMV-MVA Triplex — 5 x 108 plaque-forming unit (pfu) ±0.5 x 108 pfu of MVA Vaccine
  Arms: Vaccine Group
Biological: Placebo — 7.5% Lactose in phosphate-buffered saline [PBS]
  Arms: Placebo Group

SUMMARY:
Participants will be randomized in a 2:1 ratio to receive either two injections of CMV-MVA Triplex® or placebo administered at study Entry/Day 0 and week 4.

Vaccine Group: 60 participants will receive CMV-MVA Triplex® containing 5 x 10^8 plaque-forming unit (pfu) ±0.5 x 10^8 pfu of MVA Vaccine Encoding CMV Antigens by intramuscular (IM) deltoid injections.

Placebo Group: 30 participants will receive a volume of placebo (7.5% Lactose in phosphate-buffered saline [PBS]) that matches the volume of the active vaccine injection by IM deltoid injections.

DETAILED DESCRIPTION:
A5355 is a phase II, double-blind, randomized, placebo-controlled, multicenter study to evaluate the safety and immunogenicity of two injections of MVA Vaccine Encoding CMV antigens (Triplex®) in adults with both HIV and CMV. Participants will be randomized in a 2:1 ratio to receive either two injections of CMV-MVA Triplex® or placebo administered at study Entry/Day 0 and week 4. Participants will have follow-up visits in person or by phone for 92 weeks after the second injection, for a total of 96 weeks of follow-up. During the study, participants will have blood, urine, genital secretions, and oral secretions collected.

Enrollment will be stratified based on sex and use of gender-affirming hormones with at least 25% of participants being individuals assigned female sex at birth not on testosterone or individuals assigned male sex at birth on feminizing hormones. Special outreach to transgender and gender non-binary persons will be encouraged with exploratory stratified analysis conducted based on both gender and sex assigned at birth.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test, or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit, at any time prior to study entry, and confirmed by a licensed Western blot, or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

* Currently on continuous ART for ≥48 weeks prior to study entry. This is defined as continuous ART consisting of at least 2 nucleoside reverse transcriptase inhibitors (NRTIs) and either a protease inhibitor boosted with low dose ritonavir or with cobicistat, an integrase inhibitor, or an non-nucleoside reverse transcriptase inhibitor (NNRTI) for the 48-week period prior to study entry with no ART interruption longer than 7 consecutive days.

NOTE 1: Other ART regimens may be acceptable. For a list of acceptable ART regimens, please see the A5355 PSWP. For any regimens not listed, sites must consult the protocol team.

NOTE 2: Modifications to ART regimens prior to study entry are allowable except for the time period noted in the protocol.

* HIV-1 RNA level <75 copies/mL (or below the limit of detection of clinically certified assays) for at least 48 weeks prior to study entry, using an FDA-approved assay performed by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent. The participant must have a minimum of two values in the last 48 weeks obtained >30 days apart, with the most recent value obtained within 45 days prior to entry.

NOTE: Single determinations that are between the assay quantification limit and 500 copies/mL (i.e., "blips") are allowed as long as the preceding and subsequent determinations are both below the level of quantification. The screening value may serve as the subsequent undetectable value following a blip.

* CD4+ cell count >250 cells/μL, obtained within 45 days prior to study entry at any US laboratory that has a CLIA certification or its equivalent.
* The following laboratory values, obtained within 45 days prior to entry (unless otherwise noted) by any US laboratory that has a CLIA certification or its equivalent:

  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 75,000/mm3
  * Estimated Glomerular Filtration Rate (eGFR) >50 mL/min/1.73m2 or creatinine clearance (CrCl) >50 mL/min using the Cockcroft-Gault equation on the FSTRF website.
  * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase ≤ 3 X ULN
  * Hemoglobin A1c (HgbA1c) <6.5% (within 90 days prior to entry)
* Positive CMV immunoglobulin G antibody (IgG) serology, using an FDA-approved assay at any US laboratory that has a CLIA certification or its equivalent at any time prior to study entry.
* Participants on statin therapy must be stable on the same dose for at least the prior 12 weeks with no anticipated change in statin or dose during the first 48 weeks of study.
* For individuals of reproductive potential who are able to become pregnant, a negative serum or urine pregnancy test within 24 hours prior to study entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/CLIA-waived test.

NOTE: Individuals of reproductive potential who are able to become pregnant are defined as individuals who have reached menarche and who have not been post-menopausal for at least 12 consecutive months with follicle-stimulating hormone (FSH) ≥40 IU/mL or 24 consecutive months if an FSH is not available, i.e., who have had menses within the preceding 24 months, and have not undergone a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, or salpingectomy).

* Participants who are able to impregnate or become pregnant (i.e., of reproductive potential) and are participating in sexual activity that could lead to pregnancy must agree to practice contraception/birth control as indicated below or agree to not participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) for at least 14 days prior to the start of the 2-dose vaccine regimen at Entry/Day 0 through at least 60 days after the final vaccination at week 4.
* Individuals of reproductive potential who are able to become pregnant are defined above. Individuals of reproductive potential who are able to impregnate are defined as individuals who do not have documented azoospermia.

Acceptable contraception/birth control for this study includes the use of one or more of the following methods:

* Condoms with a spermicide
* Diaphragm or cervical cap with spermicide
* Intrauterine device (IUD)
* Hormone-based therapy (e.g., contraceptive pills, patches, implants, rings, or injections)

Participants who are not of reproductive potential are eligible without requiring the use of a contraceptive method. Acceptable documentation of lack of reproductive potential includes written documentation or oral communication from a clinician or clinician's staff in source documents of one or more of the following:

* Surgically sterile by hysterectomy, bilateral oophorectomy, or bilateral tubal ligation (documented in medical records or by ultrasound)
* Postmenopausal with participant reporting at least a 2-year history of amenorrhea or a serum follicle-stimulating hormone (FSH) >30 mIU/mL
* Surgically sterile following a successful vasectomy

NOTE: The participant may not be able to provide written proof of a partner's vasectomy, sterilization, or menopausal status, since the participant's partner is not usually enrolled in the same study to provide consent for release of this information. The verbal report from the participant of their partner's status should be written into the source documents.

* Individuals age ≥ 18 to ≤65 years at study entry.
* Ability and willingness of participant to provide informed consent.
* Willingness of participant to have study samples obtained and stored.

NOTE: Although agreement to provide genital secretion at each time-point is required for all participants, inability to produce genital secretion samples at one or more time-point is not exclusionary

Exclusion Criteria:

* Unapproved modification in ART regimen within the 12 weeks prior to study entry, or anticipated/intended modification of ART during the study period.

NOTE: Certain modifications of ART doses during the 12 weeks prior to study entry are permitted. In addition, change in formulation (e.g., from standard formulation to fixed-dose combination) is allowed within 12 weeks prior to study entry. A within-class single drug substitution (e.g., switch from nevirapine to efavirenz, from atazanavir to darunavir, from TDF to TAF) is allowed within 12 weeks prior to study entry, with the exception of a switch between any other NRTI to/from abacavir. No other changes in ART within the 12 weeks prior to study entry are permitted.

* Nadir CD4+ cell count <100 cells/μL performed by any US laboratory that has a CLIA certification or its equivalent.

NOTE: If documentation is not available, then participant recall is acceptable, subject to the referring physician's confirmation that the participant's recall is consistent with the referring physician's knowledge and judgment.

* Breastfeeding.
* History of or active autoimmune disorders, including but not limited to inflammatory bowel diseases, scleroderma, severe psoriasis, myocarditis, uveitis, pneumonitis, systemic lupus erythematosus, rheumatoid arthritis, optic neuritis, myasthenia gravis, adrenal insufficiency, untreated hypothyroidism and/or hyperthyroidism, autoimmune thyroiditis, or sarcoidosis.

NOTE: For questions related to the definition of autoimmune disorders, sites should contact the A5355 clinical management committee (CMC) per the Study Management section.

* Known allergy/sensitivity or any hypersensitivity to components of the vaccine.
* Use of anticoagulants, bleeding disorder, or condition associated with prolonged bleeding time that would contraindicate IM injection.

NOTE: Use of daily aspirin is not exclusionary.

* Use of drugs with anti-CMV activity within 14 days prior to study entry (including but not limited to ganciclovir, valganciclovir, foscarnet, cidofovir, and letermovir).

NOTE: Acyclovir and valacyclovir may be used.

* Any episode of symptomatic CMV disease within 12 months prior to study entry.
* Previous receipt at any time of any experimental CMV vaccine.
* Use of any infusion blood product or immune globulin within 3 months prior to study entry.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine, and monoclonal antibodies), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 60 days prior to study entry.

NOTE: Participants receiving stable physiologic glucocorticoid doses, defined as prednisone ≤10 mg/day or the equivalent, will not be excluded. Stable physiologic glucocorticoid doses should not be discontinued for the duration of the study. In addition, participants receiving inhaled or topical corticosteroids will not be excluded.

* Intent to use immunomodulators (e.g., IL-2, IL-12, interferons, or TNF modifiers) during the course of the study.
* Pre-existing cardiovascular disease or diabetes mellitus diagnosed by a medical provider.

NOTE 1: History of or current diagnosis of coronary artery disease, angina pectoris, myocardial infarction, previous coronary artery intervention (stenting, angioplasty), peripheral arterial disease (claudication, peripheral arterial angioplasty, or peripheral arterial bypass procedure), cerebrovascular disease (stroke or transient ischemic attack with documented carotid or aortic atherosclerosis), or abdominal aortic aneurysm are exclusionary for this study.

NOTE 2: Poorly controlled hypertension, as defined as ≥160/100 mmHg at two occasions, is exclusionary. A pre-existing history of hypertension alone is not exclusionary.

* For those >40 years of age, a 10-year American College of Cardiology/American Heart Association (ACC/AHA) cardiovascular disease (CVD) risk of >15% (http://www.cvriskcalculator.com/) within 45 days prior to study entry.
* Receipt of a vaccine within 4 weeks prior to study entry.

NOTE: These restrictions apply to any non-MVA-based vaccine, including approved and experimental SARS-Cov-2/COVID-19 vaccines.

* Receipt of MVA-based vaccines (e.g., for HIV or tuberculosis) within 1 year prior to study entry.
* Active HIV-associated dementia.
* Active hepatitis C (defined as hepatitis C virus (HCV) antibody (Ab) positive and HCV RNA detectable within 24 weeks prior to study entry).
* Active hepatitis B (defined as hepatitis B surface antibody (HBsAb) negative, hepatitis B surface antigen positive (HBsAg), and/or HBV DNA detectable within 24 weeks prior to study entry).

NOTE 1: Participants with HBV DNA suppressed on an antiviral regimen containing anti-HBV agents are eligible if they have HBV DNA BLQ within the past 24 weeks or at screening.

NOTE 2: Prior documentation of positive HBsAb is acceptable evidence that hepatitis B is not present. If HBsAb is BLQ or documentation is not available, HBsAg and HBcAb should be documented prior to study entry. Participants who have positive HBcAb but BLQ HBsAg and HBsAb (isolated HBcAb positive status) must have HBV DNA polymerase chain reaction (PCR) performed and confirmed as BLQ for participant to be eligible.

* Suspected active rectal, genital, or pharyngeal chlamydia, gonorrhea, or syphilis (based on screening test results and other clinical information). These participants need to be treated and can be rescreened 30 days or more after treatment. Treatment must be documented.

NOTE: Screening for chlamydia and gonorrhea by nucleic acid amplification test (NAAT) only. In persons with positive syphilis enzyme immunoassay (EIA) or rapid plasma regain (RPR), a treponema-based test must be performed for confirmation, however, only evidence of active infection would exclude the subject from the study.

* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness, in the opinion of the site investigator, requiring systemic treatment and/or hospitalization within 14 days prior to entry.

NOTE: See protocol for guidelines related to COVID-19 infection.

* Body temperature >38°C.
* No evidence of immunity to varicella.

NOTE: Serology should only be utilized to verify a history of varicella if the participant does not report a history of chickenpox or have documented completion of the varicella vaccine series.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of Grade ≥3 AEs | Thru week 48
Change in pp65-specific CD137+ CD8+ T cells | From Day 0 to week 12
Change in sTNFRII | Day 0 thru week 48

SECONDARY OUTCOMES:
Change in IL-6 | From day 0 to week 12, 24, 48 and 72
Change in sCD163 | From Day 0 to Weeks 12, 24, 48, 72
Change in IP-10 | From Day 0 to Weeks 12, 24, 48, 72
Change in sTNFRII | From Day 0 to Weeks 12, 24, 48, 72
Change in D-Dimers | From Day 0 to Weeks 12, 24, 48, 72
Change in IE1-specific CD137+ CD8+ T cells | From Day 0 to Week 12
Change in IE2-specific CD137+ CD8+ T cells | From day 0 to week 12
Change in pp65-specific CD137+ CD8+ T cells | From day 0 to Week 48
Change in IE1-specific CD137+ CD8+ T cells | From day 0 to Week 48
Change in IE2-specific CD137+ CD8+ T cells | From day 0 to Week 48
CMV DNA in PBMC | At weeks 12, 48, and 72
CMV DNA in urine | At weeks 12, 48, and 72
CMV DNA is genital secretion | At weeks 12,48, and 72
Viral DNA from recombinant MVA vaccine | At week 12
Occurrence of Grade ≥3 AEs | Through week 96

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gianella, MD, Study Chair — Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections
Locations (12):
- United States (12):
  - Alabama CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: With whom?
  Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  For what types of analyses?
  To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  By what mechanism will data be made available?
  Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/submit-a-proposal/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.